CLINICAL TRIAL: NCT01278446
Title: Evaluation of Hypoallergenicity of a 100% Whey, Extensively Hydrolyzed Infant Formula
Brief Title: Extensively Hydrolyzed Formula: Hypoallergenicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 09.42.PED
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Food Hypersensitivity
Keywords: Cow's Milk Allergy; CMA
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity | interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Formula (Experimental): New hydrolyzed whey formula
  Interventions: Other: Extensively hydrolyzed, whey protein infant formula
- Control Formula (Active Comparator): Commercially available hydrolyzed infant formula
  Interventions: Other: Extensively hydrolyzed, casein protein infant formula

INTERVENTIONS:
Other: Extensively hydrolyzed, whey protein infant formula — New hydrolyzed formula
  Other Names: Baby Formula
  Arms: Test Formula
Other: Extensively hydrolyzed, casein protein infant formula — Commercially available hydrolyzed infant formula
  Other Names: Baby Formula
  Arms: Control Formula

SUMMARY:
The primary objective of this clinical trial is to determine whether a new extensively hydrolyzed infant formula is hypoallergenic.

ELIGIBILITY:
Inclusion Criteria:

1. Born at term (>36 weeks gestation)
2. Two (2) months to ≤ 12 years of age at enrollment
3. Documented Cow's Milk Allergy (CMA) within the 6 months prior to enrollment by:

   1. Reported convincing allergic symptoms following an exposure to milk or a milk-containing food product and [detectable serum milk-specific IgE (>0.7 kIU/L) or positive skin prick test (wheal greater than 5 mm]), OR
   2. Physician-supervised oral food challenge that elicited immediate allergic symptoms, OR
   3. Results of laboratory tests highly predictive of clinical reactivity to milk

      * Serum milk IgE ≥15 [kIU/L]or ≥ 5 [kIU/L if younger than 1 year OR,
      * Skin prick tests mean wheal >10 mm
4. Otherwise healthy
5. If subject has asthma, atopic dermatitis, and/or rhinitis, must be well controlled
6. Expected daily intake of at least 8 oz (240 ml) of the study formula during the open challenge phase
7. Having obtained his/her legal representative's informed consent.

Exclusion Criteria:

1. Children consuming mother's milk at the time of inclusion and during the trial
2. Any chromosomal or major congenital anomalies
3. Any major gastrointestinal disease or abnormalities other than CMA
4. Chronic medical diseases (ie seizure disorders, chronic lung disease, heart problems (heart murmurs acceptable)
5. Immunodeficiency
6. Receiving free amino acid formula
7. Anti-histamine use in 7 days prior to the first food challenge (eyedrops are acceptable)
8. Oral steroid use within 14 days prior to enrollment (intranasal and topical corticosteroids are okay)
9. Unstable asthma
10. Severe uncontrolled eczema
11. Recent ( within the last 3 months) severe anaphylactic reaction to milk
12. Subject who in the Investigator's assessment cannot be expected to adhere to the study protocol
13. Currently participating in another clinical trial

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Hypoallergenicity | 14 Days
  To demonstrate that the test formula does not provoke allergenic activity

SECONDARY OUTCOMES:
Digestive Tolerance | 1 Week

CONTACTS AND LOCATIONS:
Overall Officials: Jose Saavedra, MD, Study Director — Nestle Nutrition; Anna Nowak-Wegrzyn, MD, Principal Investigator — Mount Sinai Department of Pediatrics
Locations (14):
- United States (14):
  - Little Rock Allergy & Asthma, Little Rock, Arkansas
  - Pediatric Care Medical Group, Inc, Huntington Beach, California
  - Allergy Medical Group of the North Area, Roseville, California
  - Brookstone Clinical Research Center, Columbus, Georgia
  - Aeroallergy Research Labs of Savannah, Savannah, Georgia
  - Idaho Allergy and Asthma Specialists, Eagle, Idaho
  - Deaconness Clinic, Evansville, Indiana
  - Anderson & Collins Clinical Research, Edison, New Jersey
  - Mount Sinai Faculty Practice Associates Pediatric Allergy, New York, New York
  - ENT & Allergy Associates, Newburgh, New York
  - Allergy Partners of Western North Carolina, Asheville, North Carolina
  - TTS Research, Boerne, Texas
  - Clinical Research Partners, Henrico, Virginia
  - Advanced Pediatrics, Vienna, Virginia